CLINICAL TRIAL: NCT05437835
Title: The Correlation Between the Diffusion Length of Local Anesthetics in the Subparaneural Space and Duration of Analgesia for Patients Receiving Sciatic Block
Brief Title: Diffusion Length of Local Anesthetics in the Subparaneural Space and Duration of Analgesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KYLL-2022-0490
Record Dates: First submitted 2022-06-18; First posted 2022-06-29 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Lower Extremity Fracture
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diffusion length and anesthetic effect (Experimental): diffusion length of local anesthetics in the subparaneural space could predict anesthetic effect and duration of analgesia
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — Ropivacaine 20 ml injection into the subparaneural space of sciatic nerve

SUMMARY:
Ultrasound-guided popliteal sciatic nerve block is a widely practiced technique to provide anesthesia or analgesia for below-knee surgeries. One study named the space between paraneural sheath and epimysium of sciatic nerve as the subparaneural space. It has been reported that injection into the subparaneural space has several advantages (improved the quality of the sensory block and resulted in a longer block duration) over conventional perineural injection. The investigators conducted this prospective randomized study to test the hypothesis that, during ultrasound-guided single popliteal sciatic nerve block, diffusion length of local anesthetics in the subparaneural space could predict anesthetic effect and duration of analgesia. The results of this study will develop a novel indicator to facilitate personalized medicine for patients receiving sciatic block.

DETAILED DESCRIPTION:
Introduction Below-knee surgeries are a common injury of foot, ankle and shin accompanied by severe and difficult-to-treat pain. For patients with Below-knee fractures, surgery is generally the mainstay of treatment to relieve pain and correct foot dysfunction. However, the surgical treatment can result in significant postoperative pain for at least 24 h. In addition, severe pain often leads to physical inactivity, potentially leading to hematoma, incision dehiscence or infection, thereby increasing the difficulty of postoperative nursing and the workload of medical staff. Therefore, effective postoperative analgesia is of great significance to relieve patients' pain and promote postoperative recovery.

Due to various advantages, ultrasound-guided peripheral nerve blocks have gained increasing popularity among anesthesiologists and patients. Popliteal sciatic nerve block is a widely practiced regional anesthesia technique to provide anesthesia or analgesia for below-knee surgeries because it is located superficially and is relatively easy to identify when the popliteal artery is used as an anatomical landmark. The analgesic effect of popliteal approach sciatic nerve block can just last approximately 15 hours after operation even when long-acting local anesthetics are used. But the below-knee surgeries treatment can result in significant postoperative pain for at least 24 hours. Anesthesiologists needs new ways to prolong duration times and decrease the incidence of complications.

One study named the space between paraneural sheath and epimysium of sciatic nerve as the subparaneural space. It has been reported that injection into the subparaneural space has several advantages (improved the quality of the sensory block and resulted in a longer block duration) over conventional perineural injection because paraneral sheath act as conduits for local anesthetic spread during a sciatic nerve block. However, few data are currently available in the literature evaluating analgesic effect and the diffusion length of local anesthetics in the subparaneural space for patients receiving sciatic block. To obtain more information on this topic, the investigators conducted this prospective randomized study to test the hypothesis that, during ultrasound-guided single popliteal sciatic nerve block, diffusion length of local anesthetics in the subparaneural space could predict anesthetic effect and duration of analgesia. The results of this study will develop a novel indicator to facilitate personalized medicine for patients receiving sciatic block.

Methods Subjects After obtaining approval by the Ethics Committees of the General Hospital of Ningxia Medical University (No. KYLL-2022-4940) and written informed patient consent, consecutive patients scheduled for below-knee surgery under general anesthesia combined with peripheral nerve block were enrolled in this study.

One hundred patients aged 19 to 70 years and scheduled for elective below-knee surgery under general anesthesia combined with peripheral nerve block were included. Their physical status was rated I to II by the criteria of the American Society of Anesthesiologists (ASA). Exclusion criteria were clinically significant coagulopathy, infection at the injection site, allergy to the local anesthetics, severe cardiopulmonary disease (NYHA ≥III), a body mass index > 35kg/m2, diabetic or other neuropathy, prior surgery in the popliteal region, or receiving opioids for chronic analgesic therapy. All the patients in this study received nerve block in a separate "block room" furnished with monitoring devices, drugs, and an emergency kit. These procedures were performed 30 minutes early, with the consent of patients and surgeon, because of the long preparation time and the prolonged onset time. All procedures were performed under ultrasonographic guidance (EDGE II, FUJIFILM Sonosite, USA). Eighteen-gauge intravenous access was established in the forearm in the general ward. After arrival in the block room, the investigators applied supplemental oxygen by facial mask at 5 L/min and standard monitoring (noninvasive arterial blood pressure, electrocardiography, and pulse oximetry) throughout anesthesia. Patients were premedicated with intravenous midazolam (0.02 mg/kg) and sufentanil (0.1 ug/kg). All blocks were conducted by one anesthesiologist who had substantial expertise in ultrasound-guided nerve block. The sciatic nerve block of this study was performed using a subparaneural space injection technique. When the surgical procedure involved the medial aspect of the calf and ankle, an additional ultrasound-guided femoral nerve block was performed.

1. Nerve block technique With the patient in a non-dependent lateral position, the skin was prepared with iodine and alcohol solutions. The ultrasound probe was placed transversely across the popliteal fossa at the popliteal crease. After confirming the popliteal artery, vein, and tibial nerve, the probe was moved proximally to find the bifurcation of the sciatic nerve. The neural bifurcation was identified as the point where both branches are contiguous and display a bilobular pattern. The insertion point of the needle was proximally 5 cm to the bifurcation of the sciatic nerve. A skin wheal was raised with 1mL of lidocaine 1%. Using an in-plane technique, a 22G nerve stimulation needle was advanced in parallel with the linear probe until the tip reached the subparaneural space. To confirm accurate needle tip positioning beneath the paraneural sheath, the investigators used two confirmatory steps: detecting a tactile, fascial "click" on needle passage through the paraneural sheath and observing immediate separation of the adjacent nerve and common peroneal nerve upon injection of saline (0.5mL) without neural swelling. At this point, 20 ml of 0.5% ropivacaine (AstraZeneca, Luton, UK) was injected slowly after negative blood aspiration. If neural swelling was detected under ultrasound, the needle was carefully withdrawn before resuming the injection. After ropivacaine injection, the needle was removed, and the diffusion length of local anesthetics in the paraneral sheath were measured by ultraphonic. When the surgical procedure involved the medial aspect of the calf and ankle, an additional ultrasound-guided femoral nerve block was performed. With the patient in the supine position, the femoral nerve was blocked with sterile technique using a linear probe at the middle and lower thigh. After confirming the femoral vessels, fascia iliaca, and femoral nerve, a 22G needle was inserted in-plane in a lateral-to-medial orientation and advanced toward the fascia iliaca and femoral nerve. After confirming the passage of the needle through the fascia iliaca using fascial click and a small amount of saline, the investigators injected 10 mL of 0.5% ropivacaine between the fascia iliaca and the femoral nerve. The sensory and motor blocks were evaluated every 5 minutes for 30 minutes.

   In another experiment, the investigators aim to determine the minimum effective diffusion length of local anesthetics in the subparaneural space for patients receiving sciatic block. The investigators start with 20 ml of 0.5% ropivacaine, the injection volume for the next patient was decreased by 2mL (10% of the initial volume). Conversely, if the block failed, the next patient's volume was increased by 2mL. The maximum dose used in sciatic block was limited to 25 mL of 0. 5% ropivacaine. The study plan also called for stopping after obtaining 5 consecutive successful blocks requiring less than 5 mL each, because this study was not designed to measure such small quantities.
2. Nerve block assessment After ropivacaine injection, the sensory and motor block were evaluated every 5 minutes for 30 minutes by an independent observer, who was not present during block administration and was blinded to the injected volume. Using a 23-gauge needle and cold ice, the observer assessed the sensory block in the distributions of the tibial nerve (plantar surface of the foot), deep peroneal nerve (first and second web spaces of the toes), and superficial peroneal nerve (dorsal surface of the foot). Additionally, the presence of motor blockade was tested in the tibial nerve (plantar flexion of the foot) and common peroneal nerve (dorsiflexion of the foot). The sensory and motor blockades were graded on a 4-point scale.

The block was considered a success if anesthesia and paresis were achieved within 30 minutes (a score of 3 for both sensory and motor nerves). If the blockade failed, it was classified as an incomplete block of the sensory and/or motor nerves. 30 min after nerve block, all patients received general anesthesia via the supraglottic airway. Postoperative pain was assessed using a visual analog score (VAS), in which a score of 0 indicated no pain and a score of 10 indicated the most severe pain. If the VAS was more than 4 points in the PACU, intravenous parecoxib sodium 100 mg was to be prescribed as rescue analgesia. Postoperative analgesia consisted of oral celecoxib 200 mg twice daily for 72 hours after surgery. In addition, intravenous sufentanil infusion was to be started in the PACU using a patient controlled analgesia (PCA) pump. The PCA was programmed to deliver a bolus dose of 0.5 ug/kg, without background infusion, with a lockout of 5 minutes, and a 4-hour limit of 4ug/kg.

In the first part, the primary outcome measure was the correlation between the diffusion length of local anesthetics in the subparaneural space and the duration of analgesia for patients receiving sciatic block. In the second part, the primary outcome measure was the minimum effective diffusion length of local anesthetics in the subparaneural space resulting in a successful block of the sciatic nerve in 50% of patients. The ED90 was calculated using a probit regression analysis. During the injections, any vascular punctures, paresthesias, neural swellings, or other complications were to be recorded. Three days after surgery, all patients were further interviewed by an investigator blinded to the patient doses to inquire about complications, such as persistent paresthesia and motor deficits in the block-related area. Finally, all patients were booked for a visit to the outpatient department 4 weeks postoperation for follow up by an orthopedic surgeon. The following block-related data were defined: imaging time (the time interval between contact of the US probe with the popliteal crease and the acquisition of a satisfactory picture), the needling time (the time interval between raising the skin wheal and the completion of LA injection), and the performance time (the sum of the imaging and needling times).

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective below-knee surgery under general anesthesia combined with peripheral nerve block were included. Their physical status was rated I to II by the criteria of the American Society of Anesthesiologists (ASA).

Exclusion Criteria:

* clinically significant coagulopathy, infection at the injection site, allergy to the local anesthetics, severe cardiopulmonary disease (NYHA ≥III), a body mass index > 35kg/m2, diabetic or other neuropathy, prior surgery in the popliteal region, or receiving opioids for chronic analgesic therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-07-30 (Estimated); Primary Completion 2025-07-29 (Estimated); Study Completion 2025-07-29 (Estimated)

PRIMARY OUTCOMES:
Diffusion length of ropivacaine and duration of analgesia | 3 days
  The relationship of diffusion length of 0.5% ropivacaine in the subparaneural space and duration of analgesia(sensory block time)

SECONDARY OUTCOMES:
Diffusion length of ropivacaine and duration of motor block time | 3 days
  The relationship of diffusion length of 0.5% ropivacaine in the subparaneural space and duration of motor block time

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: Undecided